CLINICAL TRIAL: NCT04900727
Title: Tobacco Control Policy-related Survey by Online Panel 2021
Brief Title: Tobacco Control Policy-related Survey 2021 (Online)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Other Study IDs: 2021 Policy Survey (Online)
Record Dates: First submitted 2021-05-17; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Survey on Tobacco Control
Keywords: Smoking; Tobacco Control Policy; Tobacco Control Measures
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Current smokers: Individuals who, at the time of the survey, smoke any forms of tobacco product either daily or occasionally.
  Interventions: Other: No intervention
- Ex-smokers: Individuals who were formerly smokers but, at the time of the survey, do not smoke at all.
  Interventions: Other: No intervention
- Never Smokers: Individuals who, at the time of the survey, have never smoked at all.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Aim: to collect further information on issues related to tobacco control which should be addressed and advocated in further tobacco control measures in Hong Kong.

The objectives of this policy-related survey by online panel are as follows:

1. to update information on prevalence of conventional cigarettes, e-cigarettes, heated tobacco products and waterpipe tobaccos;
2. to investigate the effects of new pictorial health warning policy in the public;
3. to investigate the level of public support on current and future tobacco control measures and taxation;
4. to address the timely impacts of smoke-free policies, public support for further tobacco control measures and assist COSH in shaping policy direction for government;

Current study is a repeated cross-sectional online survey based on questionnaires. A total of 2 waves of survey will be conducted 4 months apart starting from early 2021. The target sample size in each wave of survey is planned to be 900 Hong Kong residents. The online survey will be conducted by a survey agent under the monitor of applicants. All eligible registered members of the survey agent panel will be invited to respond to the questionnaire. Once a member responded to the first wave of this study, he/she would no longer receive invitation for the subsequent wave. All responses will be kept anonymously. Analysis of survey data will aim to identify current opinion on tobacco control policies and implications for future policies. All eligible subjects who complete the online survey will be included in the analysis. Comparison with past trends conducted by landline and mobile phone surveys and, where possible, extrapolation of future trends will be explored. Weightings will be applied to adjust for the sex and age of Hong Kong population, and to handle the over-sampling issues of ex- and current smokers. The data analysis will be conducted by experienced statisticians in the applicants' team.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong resident aged 15 and above
* Traditional Chinese readers

Exclusion Criteria:

* Unable to provide a consent
* Know languages other than Chinese

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Hong Kong residents
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Attitudes toward tobacco control policies | Finish all online surveys by Jan 2022
  Topics include support for future tobacco control policies (tobacco tax raise, no smoking area expansion, total ban of tobacco products), opinion on existing tobacco control policies (pictorial health warning, media advocacy).

SECONDARY OUTCOMES:
Knowledge and behaviour of smokers | Finish all online surveys by Jan 2022
  Topics include tobacco products consumption and dependence (use of product per day, time to 1st product after waking up), smoking cessation products and services (use, intention to use), influence of COVID-19 on smoking behavior (change of smoking amount), hotspot smoking (frequency of smoking in hotspots).

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Social Policy Research Limited, Hong Kong, Hong Kong